CLINICAL TRIAL: NCT03847493
Title: Analysis of Sublingual Glycocalyx Damage at ICU Admission to Predict Risk of Death - the ASGARD Study
Brief Title: Analysis of Sublingual Glycocalyx Damage at ICU Admission to Predict Risk of Death
Acronym: ASGARD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital Muenster (Other)
Responsible Party: Sponsor
Other Study IDs: ASGARD
Record Dates: First submitted 2019-02-14; First posted 2019-02-20 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-05

CONDITIONS: Sepsis; Septic Shock; Endothelial Dysfunction
Keywords: perfused boundary region; PBR; Sepsis; endothelial glycocalyx; ICU
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with suspected sepsis: Patients admitted in the ICU with the clinical suspicion of infection/sepsis.
  Interventions: Other: Endothelial Glycocalyx
- Non-sepsis Patients (control group): Patients admitted in the ICU with other conditions apart from infection/sepsis.
  Interventions: Other: Endothelial Glycocalyx

INTERVENTIONS:
Other: Endothelial Glycocalyx — Non-invasive assessment of endothelial glycocalyx dimensions.

SUMMARY:
The aim of this observative, prospective study is to evaluate if and to what extent glycocalyx damage/microcirculation data at admission in the ICU as well as during ICU stay can be predictive of mortality and clinical course in patients presenting with the suspicion of sepsis/septic shock. Therefore, the enrollment of ca 100 ICU patients is planned.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients admitted to the ICU with the clinican suspicion of sepsis/septic shock.

Exclusion Criteria:

* Underage persons, pregnant women, patients with inflammation or trauma of sublingual mucosa.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-consecutive patients admitted in the ICU of University Hospital Münster, Germany.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-04-15 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Predictive value of glycocalyx thickness regarding clinical course. | Hospital stay, an expected time of 4 weeks.
  Glycocalyx thickness measured with the use of GlycoCheck System (Perfused Boundary Region - PBR, in µm). Clinical course will be estimated with the use of e.g. Sequential Organ Failure Assessment (SOFA) score (in points).
Predictive value of glycocalyx thickness regarding mortality. | Hospital stay, an expected time of 4 weeks.
  Glycocalyx thickness measured with the use of GlycoCheck System (Perfused Boundary Region - PBR, in µm).

SECONDARY OUTCOMES:
Correlation of glycocalyx thickness with disease severity. | Hospital stay, an expected time of 4 weeks.
  Glycocalyx thickness will be measured with the use of GlycoCheck System (Perfused Boundary Region - PBR, in μm). Disease severity will be assessed with ICU scores (e.g. SOFA Score - pts)

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Kümpers, MD, Principal Investigator — University Hospital Muenster
Locations (1):
- Universitiy Hospital Muenster, Münster, Germany